CLINICAL TRIAL: NCT01557894
Title: Internet Treatment for Social Phobia in Romania: A Randomized Controlled Trial
Brief Title: Internet Treatment for Social Phobia in Romania
Acronym: iSOFIE-Ro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Tulbure Bogdan Tudor, post-doctoral researcher, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTudor
Record Dates: First submitted 2012-03-15; First posted 2012-03-20 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Phobia, Social
Keywords: Social anxiety disorders; Social phobia; Anxiety sensitivity; Irrational thinking; Guided self-help; Internet-delivered treatment
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iSOFIE (Experimental): Cognitive - Behavioral: Internet-administrated CBT for Social Phobia that contains 9 self-help text modules and exercises (i.e., behavioral experiments)
  Interventions: Other: iSOFIE
- Waitlist control group (No Intervention): Waitlist control group

INTERVENTIONS:
Other: iSOFIE — Cognitive - Behavioral: Internet-administrated CBT for social phobia that contains 9 self-help text modules and exercises (i.e., behavioral experiments)
  Arms: iSOFIE

SUMMARY:
The main aim of this study is to investigate the effectiveness of an Internet-delivered intervention for social phobia by comparing it to a waitlist control group. The second aim of the study is to track the potential changes in participants' thinking patterns. Because this is among the first guided Internet-delivered interventions conducted in Romania, the treatment credibility will also be investigated. Finally, the predictive power of anxiety sensitivity for both SAD symptoms and the treatment effectiveness will be investigated.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate the effectiveness of an internet intervention for social phobia (i.e., the iSOFIE) by comparing it to a waitlist control group. iSOFIE was derived from a previously tested program (Furmark, Holmström, Sparthan, Carlbring, & Andersson, 2006) and has been significantly shortened while retaining the most important elements. The second aim of the study is to track the potential changes in participants' thinking patterns. While this intervention is primarily based on the cognitive-behavioral model of SAD (Clark and Wells, 1995), and no specific Rational Emotive Behavior Therapy (REBT, Ellis & Dryden, 1997) will be implemented, it is hypothesized that the cognitive restructuring and exposure exercises will make participants less prone to irrational thinking (as measured by the Attitude and Belief Scale-II (ABS-II, DiGiuseppe, Leaf, Exner, & Robin, 1988). To our knowledge, no study has investigated whether an iCBT program for SAD has the potential to alter participants' irrational thinking patterns. Moreover, because this is among the first guided Internet-delivered interventions conducted in Romania, the treatment credibility of the program will be investigated. Finally, the predictive power of anxiety sensitivity for both SAD symptoms and the treatment effectiveness will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* social anxiety disorder is the primary diagnostic (according to the DSM-IV)
* access to an Internet connected computer
* be fluent in Romanian language

Exclusion Criteria:

* suicidal ideation
* ongoing psychological treatment for social anxiety disorder
* recent change in psychiatric medication (i.e., during the last 6 weeks)
* psychoses or borderline personality disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan Tudor Tulbure, post-doc, Study Director — Babes-Bolyai University, Romania; Gerhard Andersson, Professor, Study Chair — Linkoeping University
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Cluj, Romania

REFERENCES:
- [Background] Tulbure BT, Mansson KN, Andersson G. Internet treatment for social anxiety disorder in Romania: study protocol for a randomized controlled trial. Trials. 2012 Oct 30;13:202. doi: 10.1186/1745-6215-13-202. PMID 23111108
- [Derived] Tulbure BT, Szentagotai A, David O, Stefan S, Mansson KN, David D, Andersson G. Internet-delivered cognitive-behavioral therapy for social anxiety disorder in Romania: a randomized controlled trial. PLoS One. 2015 May 4;10(5):e0123997. doi: 10.1371/journal.pone.0123997. eCollection 2015. PMID 25938241
- See also: The public pages of the iSOFIE project (in Romanian) — http://www.iterapi.se/sites/isofie/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was briefly presented in various national and local newspapers, where a link to the project website (https://www.iterapi.se/sites/isofie) was provided. Interested participants registered online, read the informed consent, and filled in the screening questionnaires over the internet.
Pre-assignment Details: Of the 291 applicants 47 had high depression 35 had low social anxiety 38 could not be contacted 21 had long travel plans 10 declined participation 9 had other psychological disorders 8 were under 18 years 2 were redirected. Of the remaining 121 interviewed applicants, 66 meet the DSM-IV criteria for SAD, and 10 presented subclinical SAD symptoms.
Groups:
- Waitlist Control Group: Wait-list control group just completed a weekly social anxiety measure (LSAS-SR) for the first 9 weeks.
  Starting from week 10 these participants received the active intervention.
- iSOFIE: Cognitive - Behavioral: Internet-administrated CBT for Social Phobia that contains 9 self-help text modules and exercises (i.e., behavioral experiments)
  iSOFIE : Cognitive - Behavioral: Internet-administrated CBT for social phobia that contains 9 self-help text modules and exercises (i.e., behavioral experiments)
Period: Overall Study
Arm/Group | Waitlist Control Group | iSOFIE
Started | 38 | 38
Completed | 35 | 33
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Waitlist Control Group: Wait-list control group
- Total: Total of all reporting groups
Arm/Group | Waitlist Control Group | iSOFIE | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 38 | 76
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.85 (7.83) | 30.57 (7.96) | 28.82 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 15 | 16 | 31
Region of Enrollment [Number; unit: participants]
  Romania | 38 | 38 | 76

OUTCOME MEASURES:

1. Primary Outcome: Leibowitz Social Anxiety Scale - Self Report (LSAS-SR)
Description: The Leibowitz Social Anxiety Scale - Self Report (LSAS-SR) measures social anxiety.
  LSAS-SR presents 24 commonly anxiety-provoking situations, and asks participants to rate their fear and avoidance for each situation.
  In order to obtain the total LSAS-SR score the Anxiety and Avoidance subscales scores are added together.
  The LSAS-SR total score ranges from 0-144, with higher scores corresponding to greater social anxiety
Time Frame: pretreatment (week 0), post treatment (week 11), 6 month follow-up (week 37)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Waitlist Control Group: Wait-list control group just completed a weekly social anxiety measure (LSAS-SR) for the first 9 weeks. Starting from week 10 these participants benefited from the active intervention.
Arm/Group | Waitlist Control Group | iSOFIE
Number analyzed (Participants) | 38 | 38
units on a scale
  Pre-intervention assessment | 78.60 (16.14) | 78.47 (21.78)
  Post-intervention assessment | 73.69 (26.46) | 43.98 (23.17)
  Six month follow up | NA (NA) — Follow-up data on the waitlist control participants were not collected as this group received an active intervention starting from week 10. | 35.77 (25.44)
Statistical Analysis 1: Comparison: Waitlist Control Group vs iSOFIE; Test type: Superiority or Other; p < 0.01, ANCOVA — The a priori threshold for statistical significance was set at .05; Changes in primary outcome measures were evaluated using univariate ANCOVA, with pre-intervention scores as covariates, and group as a fixed factor

2. Primary Outcome: Social Phobia Inventory (SPIN)
Description: The Social Phobia Inventory (SPIN) is a brief (i.e., 17-item) self-report instrument measuring fear in social situations, avoidance of performance/social events, and physiological discomfort in social situations. Each item is rated on a 4-point scale.
  Thus, for SPIN the range of scores is 0-68, with higher scores reflecting higher levels of social anxiety symptomatology
Time Frame: pretreatment (week 0), post treatment (week 11), 6 month follow-up (week 37)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control Group | iSOFIE
Number analyzed (Participants) | 38 | 38
units on a scale
  Pre-intervention assessment | 45.50 (9.45) | 45.15 (9.69)
  Post-intervention assessment | 43.22 (10.94) | 27.95 (13.04)
  Six month follow up | NA (NA) — Follow-up data on the waitlist control participants were not collected as this group received an active intervention starting from week 10. | 19.74 (13.00)
Statistical Analysis 1: Comparison: Waitlist Control Group vs iSOFIE; Test type: Superiority or Other; p < 0.01, ANCOVA — The a priori threshold for statistical significance was set at .05; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Beck Depression Inventory-II (BDI-II)
Description: Beck Depression Inventory-II (BDI-II) is a 21-item self-report inventory widely used to assess DSM-IV depressive symptoms. Each item consists of four statements, scored 0-3, indicating increasing symptom severity.
  Thus, for BDI-II the range of scores is 0-63, with higher scores reflecting higher levels of depression.
Time Frame: pretreatment (week 0), post treatment (week 11), 6 month follow-up (week 37)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control Group | iSOFIE
Number analyzed (Participants) | 38 | 38
units on a scale
  Pre-intervention assessment | 15.39 (6.99) | 15.15 (7.47)
  Post-intervention assessment | 12.77 (7.27) | 7.25 (5.95)
  Six month follow up | NA (NA) — Follow-up data on the waitlist control participants were not collected as this group received an active intervention starting from week 10. | 6.44 (7.05)
Statistical Analysis 1: Comparison: Waitlist Control Group vs iSOFIE; Test type: Superiority or Other; p < 0.01, ANCOVA; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Attitude and Belief Scale-II (ABS-II)
Description: The Attitude and Belief Scale-II (ABS-II) measures rational and irrational thinking as described by Albert Ellis. The scale was designed to capture four cognitive processes (i.e., demandingness, awfulizing, low frustration tolerance, and self-downing/global evaluation) in three content areas (i.e., achievement, approval, and comfort). We selected the 72-item ABS-II because preliminary psychometrics are available for the Romanian population.
  The total ABS-II score range from 0 to 360, with higher scores corresponding to greater irrationality.
Time Frame: pretreatment (week 0), post treatment (week 11), 6 month follow-up (week 37)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control Group | iSOFIE
Number analyzed (Participants) | 38 | 38
units on a scale
  Pre-intervention assessment | 124.60 (41.50) | 120.94 (39.78)
  Post-intervention assessment | 102.51 (46.62) | 76.62 (34.81)
  Six month follow up | NA (NA) — Follow-up data on the wait-list control participants were not collected as this group received an active intervention starting from week 10. | 57.96 (31.67)
Statistical Analysis 1: Comparison: Waitlist Control Group vs iSOFIE; Test type: Superiority or Other; p < 0.01, ANCOVA

5. Secondary Outcome: Anxiety Sensitivity Index (ASI)
Description: The Anxiety Sensitivity Index (ASI) is a 16-item questionnaire that measures the beliefs about the social and somatic consequences of anxiety symptoms. The total ASI score ranges from 0 to 64, with higher scores corresponding to greater anxiety sensitivity.
Time Frame: pretreatment (week 0), post treatment (week 11), 6 month follow-up (week 37)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Waitlist Control Group | iSOFIE
Number analyzed (Participants) | 38 | 38
units on a scale
  Pre-intervention assessment | 29.00 (9.58) | 29.28 (11.40)
  Post-intervention assessment | 26.17 (10.26) | 18.38 (10.34)
  Six month follow up | NA (NA) — Follow-up data on the wait-list control participants were not collected as this group received an active intervention starting from week 10. | 13.40 (9.40)
Statistical Analysis 1: Comparison: Waitlist Control Group vs iSOFIE; Test type: Superiority or Other; p < 0.01, ANCOVA

ADVERSE EVENTS:
Arm/Group | Waitlist Control Group | iSOFIE
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 38/38 | 38/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Waitlist Control Group (N=38) | iSOFIE (N=38)
Social Anxiety (Psychiatric disorders) | 38 (38) | 38 (38) — Because assessment data were collected online Serious Adverse Events were not assessed as part of the study. Considering the inclusion criteria PI inferred that social anxiety represents Other Adverse Events that occurred in all participants.

LIMITATIONS AND CAVEATS:
1) An active control condition matched for clients' expectations, time, and therapist involvement was not included, 2)Due to personnel constrains, post-intervention SCID interviews were not blinded regarding the study conditions etc.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No